CLINICAL TRIAL: NCT01317225
Title: Use of 17α Hydroxyprogesterone Caproate for the Prevention of Preterm Labor in Patients With a Previous Episode of Threatened Preterm Labor During Current Pregnancy. Double Blind, Randomized, Controlled Trial.
Brief Title: Prevention of Preterm Labor in Patients With a Previous Episode of Threatened Preterm Labor With Progesterone
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., MD, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MHST2011-01
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Preterm Birth; Obstetric Labor, Premature
Keywords: Progesterone; Obstetric labor, premature; Short cervix
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 17 α hydroxyprogesterone caproate (Experimental): 17α-Hydroxyprogesterone caproate.
  Interventions: Drug: 17 α hydroxyprogesterone caproate
- Placebo (Placebo Comparator): Saline solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 17 α hydroxyprogesterone caproate — 250mg intramuscular (gluteal muscles) biweekly from enrollment until delivery.
  Arms: 17 α hydroxyprogesterone caproate
Drug: Placebo — 250 mg intramuscular (gluteal muscles)biweekly from enrollment until delivery.
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the use of 250 mg of intramuscular progesterone biweekly can reduce the incidence of preterm labor in patients with an episode of threatened preterm labor during the current pregnancy.

DETAILED DESCRIPTION:
Preterm birth is one of the main causes of neonatal mortality and morbidity around the world, with serious repercussions on the health system and the families of the preterm baby. Many drugs have been evaluated with the purpose of preventing preterm birth in the patient at risk. One of these drugs is 17 α hydroxyprogesterone caproate. The purpose of this study is to evaluate if the use of biweekly doses of 17 α hydroxyprogesterone caproate in patients hospitalized with the diagnosis of threatened preterm labor, defined as the presence of uterine contractions and a short cervix (below the 10th percentile for the gestational age), can reduce the incidence of preterm birth in this high risk group population.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 26 and 34 weeks of gestation.
* Cervical length (determined by transvaginal ultrasound) below the 10th percentile for the gestational age.

Exclusion Criteria:

* Multiple gestations.
* Maternal pathologies in which preterm termination of pregnancy is required.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of preterm birth (before 37 weeks of gestation) | 18 months
  Number of patients that delivered before 37 weeks of pregnancy

SECONDARY OUTCOMES:
Incidence of preterm birth before 35 weeks of pregnancy | 18 months
  To determine if the use of 17 α hydroxyprogesterone caproate can reduce the incidence of preterm birth before 35 weeks of gestation in patients with a previous episode of threatened preterm labor.
Incidence of preterm birth before 32 weeks of pregnancy | 18 months
  To determine if the use of 17 α hydroxyprogesterone caproate can reduce the incidence of preterm birth before 32 weeks of gestation in patients with a previous episode of threatened preterm labor.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo A Reyes, MD (Gyn/Ob), Principal Investigator — Saint Thomas Maternity Hospital; Rodrigo Velarde, MD (Gyn/Ob), Principal Investigator — Saint Thomas Maternity Hospital
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Provincia de Panamá, Panama